CLINICAL TRIAL: NCT02965495
Title: A Multicenter, Randomized, Double-blinded, Parallel, Placebo-controlled, Phase I/IIa Clinical Trial to Evaluate the Efficacy and Safety of Intra-articular YYD302 Once in the Treatment of Patients With Osteoarthritis of the Knee
Brief Title: Clinical Trial of YYD302 for Treatment of Osteoarthritis of the Knee
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Yooyoung Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: YY_YYD302_001/2a
Record Dates: First submitted 2016-11-02; First posted 2016-11-16 (Estimated); Last update posted 2017-12-11 (Actual); Status verified 2017-12

CONDITIONS: Osteoarthritis, Knee
Keywords: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- YYD302 2ml (Experimental): YYD302 2ml
  Interventions: Drug: YYD302 2ml
- YYD302 3ml (Experimental): YYD302 3ml
  Interventions: Drug: YYD302 3ml
- Placebo 3ml (Placebo Comparator): Phosphate buffered saline 3ml
  Interventions: Drug: Placebo 3ml

INTERVENTIONS:
Drug: YYD302 2ml — YYD302 2ml
  Arms: YYD302 2ml
Drug: YYD302 3ml — YYD302 3ml
  Arms: YYD302 3ml
Drug: Placebo 3ml — phosphate buffered saline 3ml
  Other Names: Placebo comparator 1
  Arms: Placebo 3ml

SUMMARY:
This is a multicenter, randomized, double-blinded, parallel, placebo-controlled, phase I/IIa clinical trial of YYD302 for treatment of osteoarthritis of the knee.

DETAILED DESCRIPTION:
phase I/IIa clinical trial of YYD302 for treatment of osteoarthritis of the knee

ELIGIBILITY:
Inclusion Criteria:

1. Males or Females 40 years and older
2. According to the clinical diagnosis standard of the American College of Rheumatology (ACR), someone, diagnosed as a single/both sides of osteoarthritis, who corresponds to over 3 conditions of followings.

   * Over 50 years of age
   * Less than 30 minutes of morning stiffness
   * Crepitus on active motion
   * 4 bony tenderness
   * Bony enlargement
   * Nopalpable warmth of synvium
3. Within 6 months from screening visit, someone who diagnosed with Kellgren & Lawrence Grade I~III by the radioactive examination.
4. By the Weight-bearing pain(100mm-VAS) examination, someone who has a outcome of the single or both sides of the osteoarthritis is over 40mm
5. Patient (No-responder) who has experienced steady pain in spite of dosing NSAIDs or other pain-killers in the past.
6. Patient who can walk by themselves without helper like cane or walker etc. (If the patient who has used helper routinely from previous 6 months, evaluating the patient including the helper is possible. In this case, patient needs to use same helper continuously by end of the clinical trial test.)
7. Patient who agrees to participate in this clinical trial by themselves.

Exclusion Criteria:

1. Someone who has BMI≥32kg/m² at the screening visit.
2. Patient who has an experience dosing psychoactive drug, narcotic analgesic which can have an effect on pain sense over 3 months habitually.
3. Patient who has been administrated gastrointestinal drug(for example H₂-blockers, misoprostol or proton pump inhibitors) regularly, who can't stop injecting for clinical study period.
4. Patient has attended abnormal values from screening test(2 times excess at upper limit of the normal values at ALT, AST, BUN, Serum Creatinine).
5. Patient who has rheumarthritis or other inflammatory metabolic arthritis.
6. Patients having serious gastrointestinal, liver, renal, heart disease.
7. When the inflammatory disease is occurred on joint area to patient like septic arthritis.
8. Patients having skin ailment at the injecting site of the joint region.
9. Patients having secondary osteoarthritis according to the Ochronosis, Hemochromatosis or systemic disease.
10. Patients who have severe pain like Sudek's atrophy, Paget's disease, Spinal disc herniation.
11. Poly-articular patients who have suffered seriously by osteoarthritis at other parts affect judge of the knee joint pain.
12. Patients who diagnosed clear interval disappearance at the knee joint by X-ray.
13. Patients who were administrated below drugs before baseline visit.

    * Patients who were injected HA at the target knee joint in recent 9 months.
    * Patients who were injected HA at other parts of the knee joint in recent 6 months.
    * Patients who were injected steroids into the intra-articular knee joint.
    * Patients who were administrated steroids systemically by the oral medication (But, except inhalation)
14. Patients who have joint effusion trouble were judged as a positive by tests like Patella tap test.
15. Patients who have target knee joint gotten surgical operation history including Arthroscopy within past one year (In case of having other side of knee joint or hip joint gotten surgical operation history, excepting the patients if there is possibility which can influence the target knee joint's appraisal.
16. Patients who have an operation history about target knee joint.
17. Patients who do the height weight aerobic exercise or anaerobic exercise.
18. Patients who need to be administrated anticoagulant agent together(But, except 300mg daily dose aspirin)
19. Patients who have hypersensitivity history about Investigational Product.
20. In the midst of women in their childbearing years, patients who disagree to do * contraception by medically permitted method for 12 weeks from administrating investigational product.

    * The contraception by medically permitted method: Condom, In case of using injection or insertion, In case of installing a intrauterine contraception device etc.
21. Patients who were injected other investigational product over a time within 30 days before participated in this clinical trail.
22. Besides that, the patients who have difficulty to be participated in this clinical trial continuously by Principle Investigator (PI)'s decision.

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-11; Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Rate of change of the Weight-bearing pain(100mm-VAS) on the 4, 12 weeks after administration in comparison with baseline | Change of the week 4 and 12 from baseline

SECONDARY OUTCOMES:
Rate of change of the KOOS scales on the 4, 12 weeks after administration in comparison with baseline | Week 4 and Week 12
Rate of change of the rest pain(100mm-VAS) on the 4, 12 weeks after administration in comparison with baseline | Week 4 and Week 12
Motion pain (100mm-VAS) on the 4, 12 weeks after administration in comparison with baseline | Week 4 and Week 12
Patient global assessment (100mm-VAS) on the 4, 12 weeks after administration with baseline | Week 4 and Week 12
Investigator global assessment (100mm-VAS) on the 4, 12 weeks after administration | Week 4 and Week 12
Change of the swelling in the knee joint from baseline to 4, 12 weeks after administration | Week 4 and Week 12
Change of the tenderness on pressure in the knee joint from baseline to 4, 12 weeks after administration | Week 4 and Week 12
Variation of the Range Of Motion(ROM) in the knee joint on 4, 12 weeks after administration with baseline | Week 4 and Week 12
Use of rescue medication count and the total amount on 4, 12 weeks | Week 4 and Week 12
Response rate of the Weight-bearing pain on 12 weeks in comparison with baseline | Week 12
Response rate of the OMERACT-OARSI on 12 weeks in comparison with baseline | Week 12

CONTACTS AND LOCATIONS:
Overall Officials: Chul-Won Ha, M.D, Principal Investigator — Samsung Medical Center, Department of Internal Medicine
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided